CLINICAL TRIAL: NCT06669403
Title: A Phase 1b Study to Assess the Safety, Tolerability and Pharmacokinetics of OPT101 in Patients With Community Acquired Pneumonia (CAP) With Sepsis
Brief Title: OPT101 in Patients With Community Acquired Pneumonia (CAP) With Sepsis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Op-T LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPT101-100-40
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Sepsis; Community Acquired Pneumonia (CAP)
Keywords: Sepsis; Community Acquired Pneumonia (CAP); Immunomodulator; OPT101; Op-T LLC
MeSH Terms: conditions — Sepsis; Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.9% Sodium Chloride Injection USP (Placebo Comparator): Placebo will be 50mL normal saline (Sodium Chloride), USP sterile solution provided in a 50mL pre-packaged Intravenous (IV) bag.
  Interventions: Other: Placebo
- OPT101 (Experimental): OPT101 (15-mer peptide) will be provided across 2 cohorts at 1.1 (cohort 1) and 2.8 mg/kg (cohort 2) doses . On the day of administration, the product will be diluted in saline to result in 50 mL for intravenous (IV) infusion over 120 minutes.
  Interventions: Drug: OPT101

INTERVENTIONS:
Drug: OPT101 — OPT101, is a 15-mer peptide derived from the sequence of mouse CD40L and was designed to target CD40-mediated inflammation. On the day of administration, the product will be diluted in saline to result in 50 mL for intravenous (IV) infusion over 120 minutes.
  Arms: OPT101
Other: Placebo — 0.9% Sodium Chloride Injection USP, Placebo. On the day of administration, a 50mL IV bag containing saline (0.9% Sodium Chloride Injection USP) which will serve as the placebo will be administered via intravenous (IV) infusion over 120 minutes.
  Other Names: Placebeo
  Arms: 0.9% Sodium Chloride Injection USP

SUMMARY:
OPT101-100-40 is a multicenter, randomized, placebo-controlled, multiple-ascending-dose, sequential-group, investigator- and participant-blinded, sponsor-unblinded, study of OPT101 vs placebo when administered for up to 4 days to patients admitted to the hospital for treatment of Community Acquired Pneumonia (CAP) with sepsis.

This study will be performed in patients with Community Acquired Pneumonia (CAP) with Sepsis, who are 18 years or older to evaluate the safety and tolerability of OPT101 in a population with elevated levels of pathologic CD40.

ELIGIBILITY:
Inclusion Criteria:

1. Are able and willing to give signed informed consent (legally authorized representative can provide informed consent if needed).
2. ≥18 years old;
3. Patients hospitalized for clinically suspected community acquired pneumonia (CAP), defined as the occurrence of (within 48h from hospital admission) at least 1 of the following signs:

   * respiratory rate > 30 breaths/min;
   * fever (> 38.0°C or > 100.4° F);
   * leukopenia (≤ 4,000 WBC/mm3 or leukocytosis (≥ 12,000 WBC/mm3);
   * adults ≥ 70 years of age; altered mental status with no other recognized cause;

   AND at least 1 of the following:
   * New onset of purulent sputum or change in character of sputum or increased respiratory secretions;
   * New onset or worsening cough, or dyspnea, or tachypnea;
   * Rales or bronchial breath sounds; AND Radiologic imaging (chest x-ray or CT scan) evidence of pulmonary involvement with new and persistent or progressive and persistent infiltrate, consolidation or cavitation AND SpO2 <92% at room air, or PaO2/FiO2 (or SpO2/FiO2) <300; recorded on one episode
4. Need for non-invasive supplemental oxygen (nasal cannula, simple mask, venturi or reservoir cannula/mask or heated high flow nasal cannula oxygen.
5. Females of child-bearing potential who are sexually active must not wish to get pregnant within 30 days after the end of the study and must be using at least one of the following reliable methods of contraception:

   * Hormonal contraception, systemic, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit until 30 days after the last OPT101 dose
   * A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit until 30 days after the last OPT101 dose
   * A male sexual partner who agrees to use a male condom with spermicide
   * A sterile sexual partner

Exclusion Criteria:

1. Need for endotracheal intubation and mechanical ventilation or extracorporeal membrane oxygenation (ECMO) at time of study screening
2. QTc ≥ 450 msec on screening ECG
3. Hepatic dysfunction: ALT or AST > 5 ULN; history of chronic hepatic disease (defined with Child-Pugh score ≥ 12)
4. Recent or active hepatitis A infection; test positive or have been treated for hepatitis B, hepatitis C, or HIV infection; evidence of active or untreated latent TB; a recent history of recurrent herpes zoster and/or opportunistic infection; and/or taking immunosuppressant medication.
5. Renal dysfunction: estimated glomerular filtration rate (eGFR) <50 mL/min/1.73 m2, or need for hemodialysis or hemofiltration
6. Current use of >2 immunosuppressive medications or immunosuppression status (AIDS, aplastic anemia, asplenia, systemic chemotherapy within the past 3 months, neutropenia (ANC < local LLN), solid organ or bone marrow transplant recipients)
7. Treatment with prohibited medication within 5 half-lives, and inability to stop during treatment period
8. Anticipated discharge from the hospital or transfer to another hospital within 48 hours of screening
9. Allergy to OPT101or any component of OPT101 formulation
10. Participation in other interventional clinical trials
11. Pregnancy:

    * positive or missing pregnancy test before first drug intake or day 1
    * pregnant or lactating women;
    * Women of childbearing potential and fertile men who do not agree to use at least one primary form of contraception for the duration of the study
12. Current hospital stay >72h
13. Complicated CAP-associated conditions, such as fungal pulmonary infection, tuberculosis infection, abscess, empyema, significant bilateral pleural effusion, massive pulmonary embolism
14. Weight is over 250lbs
15. Any other condition which the Principal Investigator feels may jeopardize the safety of the patient or the objectives of the study. The Principal Investigator should make this determination in consideration of the patient's medical history and current clinical condition.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 30 days
  Treatment emergent adverse events will be recorded and assessed by CTCAE v4.0
Incidence of serious adverse events (SAEs) | 30 days
  SAEs will be recorded and assessed by CTCAE v4.0
Incidence of TEAEs leading to study drug discontinuation | 30 days
Incidence and characteristics of presumed infusion reactions | 30 days
  Recorded as an adverse event

SECONDARY OUTCOMES:
To measure the serum pharmacokinetics of OPT101 | 30 days
  Serum concentrations of OPT101 to determine AUCO-24
To measure the serum pharmacokinetics of OPT101 | 30 days
  Serum concentrations of OPT101 to determine Cmax
To measure the serum pharmacokinetics of OPT101 | 30 days
  Serum concentrations of OPT101 to determine Tmax
To measure the serum pharmacokinetics of OPT101 | 30 days
  Serum concentrations of OPT101 to determine t1/2
To measure the serum pharmacokinetics of OPT101 | 30 days
  Serum concentrations of OPT101 to determine Vz/F

OTHER OUTCOMES:
To observe the changes in degree of sepsis via Pneumonia Severity Index (PSI) | 30 days
  Pneumonia Severity Index (PSI) predicts the need for hospitalization for people with Community Acquired Pneumonia (CAP). Patients are ranked by Risk Class (I , II, III, IV or V). Patients with CAP categorized as Risk Class of I and II can be treated at home. Patients with CAP categorized as Risk Class III may be treated at home or may require a short hospital stay. Patients with CAP categorized as Risk Class of IV and V require hospitalization.
To observe the changes in degree of sepsis via Sequential Organ Failure Assessment (SOFA) score | 30 days
  SOFA grading, minimum value is 0 (normal) and maximum value is 4 (highest degree of dysfunction/failure). The higher the score, the worse the outcome.
To observe the changes in degree of sepsis via Cytokine Release Syndrome (CRS) grading | 30 days
  CRS is graded from Grade 1 to Grade 4. Grade 1 is the best outcome and Grade 4 is the worst outcome in terms of change in degree of sepsis. CRS parameters used for grading include fever, hypotension and hypoxia.
Evaluate Pharmacodynamic Effects of OPT101 | 30 days
  Quantitation of Th40 to Treg ratio
Evaluate Pharmacodynamic Effects of OPT101 | 30 days
  Quantitation of peripheral blood B cells
Evaluate Pharmacodynamic Effects of OPT101 | 30 days
  Quantitation of macrophages
Evaluate Pharmacodynamic Effects of OPT101 | 30 days
  Quantitation inflammatory biomarkers
Evaluate Pharmacodynamic Effects of OPT101 | 30 days
  Quantitation of Th40 cells,

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD FAAAAI, Study Director
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No